CLINICAL TRIAL: NCT02388984
Title: A Randomized, Double Blind, Multi-Center Study of Compound Danshen Dripping Pills in Patients With Diabetic Retinopathy (Syndrome Of Qi-Stagnation and Blood Stasis)
Brief Title: Phase III Study of Compound Danshen Dripping Pills to Treat Diabetic Retinopathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM9001-04
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Non-proliferative Diabetic Retinopathy
MeSH Terms: interventions — T89 herbal drug

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compound danshen dripping pills (Experimental): Compound danshen dripping pills,20pills,tid. Duration: 24 weeks.
  Interventions: Drug: Compound danshen dripping pills
- Placebo (Placebo Comparator): Placebo,20pills,tid. Duration: 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Compound danshen dripping pills — Dosage form:pill. Dosage:20pills. Frequency:three times per day. Duration:24 weeks.
  Other Names: Dantonic®
  Arms: Compound danshen dripping pills
Drug: Placebo — Dosage form:pill. Dosage:20pills. Frequency:three times per day. Duration:24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Compound Danshen Dripping Pills in patients with diabetic retinopathy(Syndrome Of Qi-Stagnation and Blood Stasis).

DETAILED DESCRIPTION:
Compound danshen dripping pills is a kind of traditional Chinese medicine(TCM), consists of Danshen (Radix Salviae Miltiorrhizae), Sanqi (Radix Notoginseng) and borneol. This study is being conducted to evaluate the efficacy and safety of compound danshen dripping pills in patients with diabetic retinopathy(Syndrome Of Qi-Stagnation and Blood Stasis), when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with non-proliferative diabetic retinopathy(NPDR) and TCM syndrome differentiation of qi-stagnation and blood stasis.
2. aged 30-70 years
3. voluntary signs the informed consent

One eye met the inclusion criteria can be used as research object, if both eyes met the inclusion criteria, please record respectively, and select one eye for efficacy evaluation with reference to the following principles:

When the two eyes of fundus conditions in different clinical stage, choose the more serious one.

When the two eyes of fundus conditions in the same clinical stage, choose the eye easier for clinical operation.

Exclusion Criteria:

1. HbAlc>8%, sustained hyperglycemia.
2. The patients who have been received the therapy of Retina laser photocoagulation or diagnosed with proliferative diabetic retinopathy (one or two eyes).
3. Diabetic retinopathy caused by type 1 diabetes mellitus.
4. Combined with glaucoma, uveitis, ocular neuropathy and severe cataract etc.
5. Combined with primarily severe diseases such as cardiovascular, hepatic，renal illness , hemopoietic system disease, and psychosis. Serum transaminase is higher than the limit of normal value of 1.5 times.
6. Diabetic nephropathy with renal failure (Azotemia or Uremia).
7. For women of child-bearing potential: pregnant or lactating or intending to become pregnant. Having any allergic reaction to some drugs.
8. Participated in other clinical trial within 3 months.
9. Used drugs for the treatment of diabetic retinopathy within 1 week.
10. Blood pressure > 160/100 (systolic above 160 or diastolic above 100).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The total effective rate of Fundus changes, the severity of diabetic retinopathy change from baseline at the end of week 24 compared to placebo | 24weeks

SECONDARY OUTCOMES:
Symptoms scores of TCM change from baseline at the end of week 24 compared to placebo | 24 weeks.
Corrected visual acuity change from baseline at the end of week 24 compared to placebo | 24 weeks.
The severity of macular edema change from baseline at the end of week 24 compared to placebo | 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Study Director — Tasly Group, Co. Ltd.
Locations (16):
- China (16):
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Dongfang Hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Southwest Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Institute of Ophthalmology, Zhengzhou, Henan
  - Hubei Provincial Hospital of TCM, Wuhan, Hubei
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Jiangsu Province Hospital of TCM, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Shenyang He Eye Hospital, Shenyang, Liaoning
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Teaching Hospital of Chengdu University of TCM, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No